CLINICAL TRIAL: NCT00930800
Title: The Effect of Exercise Training on Exercise Capacity, Physical Activity, and Health-related Quality of Life in Children After Repair of Congenital Heart Defect
Brief Title: Exercise Training in Children With Congenital Heart Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200712010R
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Congenital Heart Disease
Keywords: Exercise capacity; Physical activity; Quality of life
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Other): Dance Dance Revolution (DDR)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Using a video game so-called Dance Dance Revolution (DDR)
  Other Names: Dance Dance Revolution (DDR)

SUMMARY:
The purpose of this study was to investigate the effects of exercise training on exercise capacity, physical activity (PA), health-related quality of life (HRQoL), and the psychosocial factors affecting PA in sedentary congenital heart defect (CHD) children and healthy sedentary children. The degree of improvement after exercise training were compared between CHD children and healthy sedentary children.

DETAILED DESCRIPTION:
Exercise groups took 12-week exercise training, twice in hospital and once at home, using a video game so-called Dance Dance Revolution (DDR), while the control group kept their daily routines.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital heart defect s/p repair > 6 months
* Sedentary lifestyle

Exclusion Criteria:

* Unstable hemodynamics
* Impaired mental and cognition
* Systemic disease

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
maximal treadmill exercise test | 12 wks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan